CLINICAL TRIAL: NCT03263884
Title: Repetitive Transcranial Magnetic Stimulation and the Development of Ongoing Muscle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Medical Doctor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20170041
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Pain Relief
Keywords: nerve growth factor; repetitive transcranial magnetic stimulation; dorsolateral prefrontal cortex
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real treatment group (Experimental): Transcranial magnetic stimulation (TMS) is used to stimulate small regions of the brain. During a TMS procedure, a magnetic field generator, or "coil", is placed near the head of the person receiving the treatment. The coil produces small electric currents in the region of the brain just under the coil via electromagnetic induction.
  The protocol used in this research includes 20 minutes of 10Hz stimulation, 5 seconds on, 10 seconds off, at 110% RMT, for a total of 4000 pulses.
  Interventions: Device: Repetitive trancranial magnetic stimulation (rTMS) group
- Sham treatment group (Sham Comparator): Sham coil is used to mimic the clicking sound of the TMS coil and skin stimulation
  Interventions: Device: Sham group

INTERVENTIONS:
Device: Repetitive trancranial magnetic stimulation (rTMS) group — Repetitive trancranial magnetic stimulation is applied on the dorsolateral prefrontal cortex. The protocol consists on 20 minutes of 10Hz stimulation, 5 seconds on, 10 seconds off, at 110% RMT, for a total of 4000 pulses.
  Arms: Real treatment group
Device: Sham group — A sham coil is used to mimic the clicking sound of the trancranial magnetic coil and skin stimulation.
  Arms: Sham treatment group

SUMMARY:
The main purpose of the study is to assess the mechanisms of repeated sessions of repetitive trancranial magnetic stimulation (rTMS) applied on left dorsolateral prefrontal cortex on the development of pain in a prolonged muscle pain model.

DETAILED DESCRIPTION:
This study aims to investigate whether i) rTMS of left DLPFC will reduce the severity and duration of experimentally induced muscle pain when a 5-day course of treatment is given immediately following an initial nerve growth factor (NGF) injection; ii) the analgesic effects of left DLPFC rTMS will be related to an improved cognitive network function as assessed by electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Speak and understand English.

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Previous experience with rTMS
* Contraindications to rTMS application (history of epilepsy, metal in the head or jaw etc.).
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Pain relief | Change from baseline at 2 weeks
  Pain on an 11-point numerical rating scale (0 = no pain, 10 = most intense pain imaginable)

SECONDARY OUTCOMES:
Muscle soreness | Change from baseline at 2 weeks
  7-point Likert scale; 0 = 'a complete absence of soreness', 1 = 'a light soreness in the muscle felt only when touched/vague ache', 2 = 'a moderate soreness felt only when touched/a slight persistent ache', '3 = 'a light muscle soreness when lifting or carrying objects', 4 = 'a light muscle soreness, stiffness or weakness when moving the wrist without gripping an object', 5 = 'a moderate muscle soreness, stiffness or weakness when moving the wrist', 6 = 'a severe muscle soreness, stiffness or weakness that limits the ability to move'
Patient-rated Tennis Elbow Evaluation | Change from baseline at 2 weeks
  The Patient-rated Tennis Elbow Evaluation will be used to assess average pain and disability of the injected arm
Attention network test | Change from baseline at 2 weeks
  This task assesses cognitive function in 3 domains: alerting, orienting, and executive function
Pressure pain thresholds | Change from baseline at 2 weeks
  Pressure applied to the surface of the skin using a handheld algometer.
Cuff pressure algometry | Change from baseline at 2 weeks
  The experimental setup consists of a tourniquet cuff, a computer-controlled air compressor and an electronic visual analog scale VAS (Aalborg University, Denmark). The cuff is connected to the compressor and wrapped around the leg. The pain intensity is recorded with the electronic VAS and sampled at 10 Hz. The "0 cm" and "10 cm" extremes on the VAS are defined as "no pain" and as "maximal pain", respectively. The compression rate of the cuff is programmed on and controlled by a computer.
EEG recordings | Change from baseline at 1 weeks
  we will record brain activity in the following conditions: eyes closed rest, performance of a computer-based cognitive task (ANT).

CONTACTS AND LOCATIONS:
Overall Officials: Enrico De Martino, MD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No